CLINICAL TRIAL: NCT03173586
Title: Association Between Sugar Sweetened Beverage Intake and Biomarkers of Cardiometabolic Risk in US Women
Brief Title: Sugar Sweetened Beverage Intake and Biomarkers of Cardiometabolic Risk in US Women
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Vasanti Malik, Research Scientist, Harvard School of Public Health (HSPH)
Other Study IDs: 1999-P-011114
Record Dates: First submitted 2017-05-26; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Biomarkers
Keywords: Sugar sweetened beverage, biomarker
MeSH Terms: interventions — Sugar-Sweetened Beverages; Artificially Sweetened Beverages; 5-Aminolevulinate Synthetase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The major goal of the project was to analyze blood samples collected from 33,000 women participating in the Nurses' Health Study. The aim of the original grant was to asses plasma sex hormone levels in relation to risk of breast cancer; plasma beta-carotene, Vitamin E and omega-3 fatty acids and risk of breast and colon cancer; specific lipoprotein fractions, apoproteins and fatty acids and risk of CVD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NHS: Least-squares mean (95% CI) concentrations of biomarkers by frequency of sugar sweetened beverage (SSB) intake among participants free of diabetes and cardiovascular disease in the NHS.
  Least-squares mean (95% CI) concentrations of biomarkers by frequency of artificially sweetened beverage (ASB) intake among participants free of diabetes and cardiovascular disease in the NHS.
  Least-squares mean (95% CI) concentrations of biomarkers by frequency of fruit juice intake among participants free of diabetes and cardiovascular disease in the NHS.
  Interventions: Other: Sugar sweetened beverage (SSB)

INTERVENTIONS:
Other: Sugar sweetened beverage (SSB) — This is an observational study examining sugar sweetened beverage intake in relation to biomarkers in the NHS.
  Other Names: Artificially sweetened beverage (ASB), juice

SUMMARY:
This study is a secondary analysis of data collected in the Nurses' Health Study (NHS) that will evaluat the association between intake of sugar sweetened beverages (SSB), juice and artificially sweetened beverages in relation to biomarkers of hepatic function, lipid metabolism, inflammation and glycemic control.

DETAILED DESCRIPTION:
The investigators will analyze cross-sectional data from 8,492 participants in the Nurses' Health Study who were free of diabetes and cardiovascular disease to evaluate the association between intake of sugar sweetened beverages (SSB), juice and artificially sweetened beverages (ASB) and biomarkers of hepatic function, lipid metabolism, inflammation and glycemic control. Biomarkers were measured from blood samples that were collected in 2 cycles, approximately 10 years apart.

Specifically, multivariate linear regression will be used to assess the associations of SSB, ASB, and fruit juice intake with concentrations of fetuin-A, alanine transaminase, gamma-glutamyl transferase, triglycerides, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), total cholesterol, C-reactive protein (CRP), intracellular adhesion molecule 1 (ICAM-1), vascular cell adhesion protein 1 (VCAM-1), adiponectin, insulin, and hemoglobin A1c as well as total cholesterol/HDL-C ratio.

ELIGIBILITY:
Inclusion Criteria:

For the current study, we included participants who provided a blood sample and were previously selected as controls for nested case-control analyses of type 2 diabetes, coronary heart disease, stroke, colon cancer, colon polyps, pancreatic cancer, and breast cancer in the Nurse's Health Study.

Exclusion Criteria:

Participants with self-reported prevalent diabetes or cardiovascular disease (CVD) at blood draw were excluded. After exclusions, a total of 8,492 individuals (6,961 from cycle 1 and 1,531 from cycle 2) with valid beverage intake data were included in the current analysis.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Our analysis was based on a cohort of female registered nurses.
Study Population: The Nurses' Health Study (NHS) is a prospective cohort study of 121,700 female registered nurses aged 30-55 years at baseline in 1976. Mailed questionnaires were administered biennially to collect data on medical, dietary, and lifestyle factors, with a follow-up rate exceeding 90% for each 2-year cycle. Blood samples were collected from 32,826 participants between 1989 and 1990 (biospecimen collection cycle 1) and 18,717 participants between 2000 and 2001 (biospecimen collection cycle 2). Participants who provided a blood specimen were generally similar to those who did not in terms of diet and lifestyle
Sampling Method: Non-Probability Sample
Enrollment: 33000 (Actual)
Dates: Start 1999-09-16 (Actual); Primary Completion 2009-03-31 (Actual); Study Completion 2009-03-31 (Actual)

PRIMARY OUTCOMES:
Fetuin-A | Blood collection cycle 1 (1989-1990)
  Biomarkers of liver function
Fetuin-A | Blood collection cyle 2 (2000-2001)
  Biomarkers of liver function
Alanine transaminase | Blood collection cycle 1 (1989-1990)
  Biomarkers of liver function
Alanine transaminase | Blood collection cyle 2 (2000-2001)
  Biomarkers of liver function
Gamma-glutamyl transferase | Blood collection cycle 1 (1989-1990)
  Biomarkers of liver function
Gamma-glutamyl transferase | Blood collection cyle 2 (2000-2001)
  Biomarkers of liver function

SECONDARY OUTCOMES:
Triglycerides | Blood collection cycle 1 (1989-1990)
  Biomarkers of lipid metabolism
Triglycerides | Blood collection cycle 2 (2000-2001)
  Biomarkers of lipid metabolism
High-density lipoprotein cholesterol (HDL-C) | Blood collection cycle 1 (1989-1990)
  Biomarkers of lipid metabolism
High-density lipoprotein cholesterol (HDL-C) | Blood collection cycle 2 (2000-2001)
  Biomarkers of lipid metabolism
Low-density lipoprotein cholesterol (LDL-C) | Blood collection cycle 1 (1989-1990)
  Biomarkers of lipid metabolism
Low-density lipoprotein cholesterol (LDL-C) | Blood collection cycle 2 (2000-2001)
  Biomarkers of lipid metabolism
Total cholesterol | Blood collection cycle 1 (1989-1990)
  Biomarkers of lipid metabolism
Total cholesterol | Blood collection cycle 2 (2000-2001)
  Biomarkers of lipid metabolism
Total cholesterol/HDL-C ratio | Blood collection cycle 1 (1989-1990)
  Biomarkers of lipid metabolism
Total cholesterol/HDL-C ratio | Blood collection cycle 2 (2000-2001)
  Biomarkers of lipid metabolism
C-reactive protein (CRP) | Blood collection cycle 1 (1989-1990)
  Biomarkers of inflammation
C-reactive protein (CRP) | Blood collection cycle 2 (2000-2001)
  Biomarkers of inflammation
Intracellular adhesion molecule 1 (ICAM-1) | Blood collection cycle 1 (1989-1990)
  Biomarkers of inflammation
Intracellular adhesion molecule 1 (ICAM-1) | Blood collection cycle 2 (2000-2001)
  Biomarkers of inflammation
Vascular cell adhesion protein 1 (VCAM-1) | Blood collection cycle 1 (1989-1990)
  Biomarkers of inflammation
Vascular cell adhesion protein 1 (VCAM-1) | Blood collection cycle 2 (2000-2001)
  Biomarkers of inflammation
Insulin | Blood collection cycle 1 (1989-1990)
  Biomarkers of glucose metabolism
Insulin | Blood collection cycle 2 (2000-2001)
  Biomarkers of glucose metabolism
Hemoglobin A1c | Blood collection cycle 1 (1989-1990)
  Biomarkers of glucose metabolism
Hemoglobin A1c | Blood collection cycle 2 (2000-2001)
  Biomarkers of glucose metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Vasanti Malik, ScD, Principal Investigator — Research Scientist
Locations (1):
- Harvard T.H. Chan School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data are de-identified

REFERENCES:
- [Background] Malik VS, Popkin BM, Bray GA, Despres JP, Willett WC, Hu FB. Sugar-sweetened beverages and risk of metabolic syndrome and type 2 diabetes: a meta-analysis. Diabetes Care. 2010 Nov;33(11):2477-83. doi: 10.2337/dc10-1079. Epub 2010 Aug 6. PMID 20693348
- [Background] Xi B, Huang Y, Reilly KH, Li S, Zheng R, Barrio-Lopez MT, Martinez-Gonzalez MA, Zhou D. Sugar-sweetened beverages and risk of hypertension and CVD: a dose-response meta-analysis. Br J Nutr. 2015 Mar 14;113(5):709-17. doi: 10.1017/S0007114514004383. Epub 2015 Mar 4. PMID 25735740
- [Background] de Koning L, Malik VS, Kellogg MD, Rimm EB, Willett WC, Hu FB. Sweetened beverage consumption, incident coronary heart disease, and biomarkers of risk in men. Circulation. 2012 Apr 10;125(14):1735-41, S1. doi: 10.1161/CIRCULATIONAHA.111.067017. Epub 2012 Mar 12. PMID 22412070
- [Background] Bazzano LA, Li TY, Joshipura KJ, Hu FB. Intake of fruit, vegetables, and fruit juices and risk of diabetes in women. Diabetes Care. 2008 Jul;31(7):1311-7. doi: 10.2337/dc08-0080. Epub 2008 Apr 4. PMID 18390796
- [Background] Schulze MB, Manson JE, Ludwig DS, Colditz GA, Stampfer MJ, Willett WC, Hu FB. Sugar-sweetened beverages, weight gain, and incidence of type 2 diabetes in young and middle-aged women. JAMA. 2004 Aug 25;292(8):927-34. doi: 10.1001/jama.292.8.927. PMID 15328324
- [Background] Nettleton JA, Lutsey PL, Wang Y, Lima JA, Michos ED, Jacobs DR Jr. Diet soda intake and risk of incident metabolic syndrome and type 2 diabetes in the Multi-Ethnic Study of Atherosclerosis (MESA). Diabetes Care. 2009 Apr;32(4):688-94. doi: 10.2337/dc08-1799. Epub 2009 Jan 16. PMID 19151203
- [Background] de Koning L, Malik VS, Rimm EB, Willett WC, Hu FB. Sugar-sweetened and artificially sweetened beverage consumption and risk of type 2 diabetes in men. Am J Clin Nutr. 2011 Jun;93(6):1321-7. doi: 10.3945/ajcn.110.007922. Epub 2011 Mar 23. PMID 21430119
- [Background] Willett WC, Sampson L, Stampfer MJ, Rosner B, Bain C, Witschi J, Hennekens CH, Speizer FE. Reproducibility and validity of a semiquantitative food frequency questionnaire. Am J Epidemiol. 1985 Jul;122(1):51-65. doi: 10.1093/oxfordjournals.aje.a114086. PMID 4014201
- [Background] Salvini S, Hunter DJ, Sampson L, Stampfer MJ, Colditz GA, Rosner B, Willett WC. Food-based validation of a dietary questionnaire: the effects of week-to-week variation in food consumption. Int J Epidemiol. 1989 Dec;18(4):858-67. doi: 10.1093/ije/18.4.858. PMID 2621022
- [Background] Ley SH, Sun Q, Jimenez MC, Rexrode KM, Manson JE, Jensen MK, Rimm EB, Hu FB. Association between alcohol consumption and plasma fetuin-A and its contribution to incident type 2 diabetes in women. Diabetologia. 2014 Jan;57(1):93-101. doi: 10.1007/s00125-013-3077-8. Epub 2013 Oct 9. PMID 24105100
- [Background] Nimptsch K, Brand-Miller JC, Franz M, Sampson L, Willett WC, Giovannucci E. Dietary insulin index and insulin load in relation to biomarkers of glycemic control, plasma lipids, and inflammation markers. Am J Clin Nutr. 2011 Jul;94(1):182-90. doi: 10.3945/ajcn.110.009555. Epub 2011 May 4. PMID 21543531
- [Background] Sun Q, Cornelis MC, Manson JE, Hu FB. Plasma levels of fetuin-A and hepatic enzymes and risk of type 2 diabetes in women in the U.S. Diabetes. 2013 Jan;62(1):49-55. doi: 10.2337/db12-0372. Epub 2012 Aug 24. PMID 22923470
- [Background] Malik VS, Pan A, Willett WC, Hu FB. Sugar-sweetened beverages and weight gain in children and adults: a systematic review and meta-analysis. Am J Clin Nutr. 2013 Oct;98(4):1084-102. doi: 10.3945/ajcn.113.058362. Epub 2013 Aug 21. PMID 23966427
- [Background] Liu S, Manson JE, Buring JE, Stampfer MJ, Willett WC, Ridker PM. Relation between a diet with a high glycemic load and plasma concentrations of high-sensitivity C-reactive protein in middle-aged women. Am J Clin Nutr. 2002 Mar;75(3):492-8. doi: 10.1093/ajcn/75.3.492. PMID 11864854
- [Background] Fung TT, Malik V, Rexrode KM, Manson JE, Willett WC, Hu FB. Sweetened beverage consumption and risk of coronary heart disease in women. Am J Clin Nutr. 2009 Apr;89(4):1037-42. doi: 10.3945/ajcn.2008.27140. Epub 2009 Feb 11. PMID 19211821
- [Background] Pan A, Malik VS, Schulze MB, Manson JE, Willett WC, Hu FB. Plain-water intake and risk of type 2 diabetes in young and middle-aged women. Am J Clin Nutr. 2012 Jun;95(6):1454-60. doi: 10.3945/ajcn.111.032698. Epub 2012 May 2. PMID 22552035
- [Background] Pan A, Malik VS, Hao T, Willett WC, Mozaffarian D, Hu FB. Changes in water and beverage intake and long-term weight changes: results from three prospective cohort studies. Int J Obes (Lond). 2013 Oct;37(10):1378-85. doi: 10.1038/ijo.2012.225. Epub 2013 Jan 15. PMID 23318721
- [Background] Malik VS, Chiuve SE, Campos H, Rimm EB, Mozaffarian D, Hu FB, Sun Q. Circulating Very-Long-Chain Saturated Fatty Acids and Incident Coronary Heart Disease in US Men and Women. Circulation. 2015 Jul 28;132(4):260-8. doi: 10.1161/CIRCULATIONAHA.114.014911. Epub 2015 Jun 5. PMID 26048094
- [Background] AlEssa HB, Ley SH, Rosner B, Malik VS, Willett WC, Campos H, Hu FB. High Fiber and Low Starch Intakes Are Associated with Circulating Intermediate Biomarkers of Type 2 Diabetes among Women. J Nutr. 2016 Feb;146(2):306-17. doi: 10.3945/jn.115.219915. Epub 2016 Jan 13. PMID 26764316
- [Background] Yu Z, Malik VS, Keum N, Hu FB, Giovannucci EL, Stampfer MJ, Willett WC, Fuchs CS, Bao Y. Associations between nut consumption and inflammatory biomarkers. Am J Clin Nutr. 2016 Sep;104(3):722-8. doi: 10.3945/ajcn.116.134205. Epub 2016 Jul 27. PMID 27465378